CLINICAL TRIAL: NCT01493583
Title: Central Nervous Processing of Visual Food Stimuli in Severely Obese Subjects and After Roux-en Y Gastric Bypass Surgery - a FMRI Study
Brief Title: Central Nervous Processing of Visual Food Stimuli in Severely Obese Subjects
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Competence Network for Adiposity funded by the German Federal Ministry of Education and Research (FKZ: 01GI0837) and (FKZ: 01GI0849) (Unknown)
Responsible Party: Principal Investigator, Bernd Schultes, Prof. Dr. med., Cantonal Hospital of St. Gallen
Other Study IDs: EKSG09/033/2B; 09/033/2B (Other: ID by EKSG)
Record Dates: First submitted 2011-12-02; First posted 2011-12-16 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2013-03

CONDITIONS: Obesity
Keywords: severely obese; Roux-en Y gastric bypass surgery (RYGB); brain activity by fMRI; visual presentation of food and non-food-related pictures
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- severely obese women
- Women after Roux-en Y gastric bypass surgery: Women recruited for this group had undergone Roux-en Y gastric bypass surgery at least one year before. In this women measurement of brain activity and gastrointestinal and metabolic response took place between 13 and 106 month after surgery.
- lean women

SUMMARY:
Recent evidence has pointed to distinct alterations of brain functions in obese subjects some of which may even be causative for their obesity. The objective of this study was to examine food and non food related alterations in brain functions after excessive weight loss due to Roux-en Y gastric bypass surgery (RYGB), one of the most successful therapeutic approaches for long lasting weight loss. The investigators hypothesized that obese as compared with lean women show an altered activation pattern in the brain areas involved in the homeostatic regulation of eating behavior, i.e. the hypothalamus, in reward-related brain areas, such as the orbital frontal cortex (OFC) and the striatum as well as in prefrontal inhibitory control areas. Furthermore, the investigators hypothesized that women who had undergone a RYGB operation show a brain activity pattern that more closely mimics that of lean than severely obese women. In a supplementary test the investigators will assess gastrointestinal and metabolic response to a standardized meal in order to elucidate putative correlation of these responses with the results of fMRI scannings.

ELIGIBILITY:
Inclusion Criteria:

* women with BMI > 35kg/m2
* women, who had undergone gastric bypass surgery at least one year ago
* lean women

Exclusion Criteria:

* known psychiatric or neurological diseases
* current medication with drug acting on the central nervous system
* drugs that are known to affect eating behavior
* contraindication for the fMRI scanning, e.g. metal implants or metal containing tattoos

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely obese (body mass index; BMI > 35 kg/m2) women and previously severely obese women who had undergone a Roux-en Y gastric bypass operation were recruited from the Interdisciplinary Obesity Center, cantonal hospital St. Gallen (Switzerland), and the adiposity platform of the University of Tübingen.
  lean control women were recruited in St. Gallen and in Tübingen
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
brain activity | brain activity was measured at a single time point in all three groups; of note: women after Roux-en Y gastric bypass surgery were measured between 13 and 106 month after surgery.
  In all women brain activity was assessed by functional magnetic resonance imaging (fMRI, BOLD Method, 1.5 Tesla fMRI Scanner, Siemens, Erlangen, Germany) during the presentation of food and non-food related pictures as well as during state conditions.
  In all three groups, brain activity was measured at a single time point. Of note, women, who had undergone Roux-en Y gastric bypass surgery were measured between 13 and 106 month after surgery. Brain activity was not measured before surgery in this group.

SECONDARY OUTCOMES:
gastrointestinal and metabolic responses to standardized meal | measured at a single time point in all three groups; of note: women after Roux-en Y gastric bypass surgery were measured between 13 and 106 month after surgery at a single time point
  The gastrointestinal and metabolic responses to standardized meal were measured in the morning between 7:30 and 10:30 a.m.
  gastrointestinal and metabolic response were measured in all women at a single time point. Of note, women, who had undergone Roux-en Y gastric bypass surgery were measured between 13 and 106 month after surgery. Gastrointestinal and metabolic responses were not measured before surgery in this group.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Schultes, Prof. Dr. med., Principal Investigator — Interdisciplinary Obesity Center, Kantonal Hospital St. Gallen, Rorschach, Switzerland; Niels Birbaumer, Prof. Dr., Principal Investigator — Institute of Medical Psychology and Behavioural Neurobiology, University of Tübingen, Tübingen, Germany
Locations (1):
- Interdisciplinary Obesity Center, Cantonal Hospital St. Gallen, Rorschach, Switzerland